CLINICAL TRIAL: NCT02242136
Title: Formation, Orientation and Rehabilitation by Means of Narrative Exposure Therapy (FORNET) for Returning Soldiers of the African Union Mission to Somalia, Male and Female Ex-combatants in Burundi
Brief Title: Treatment of Posttraumatic Stress Disorder and Aggressive Behavior in Soldiers and Ex-combatants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Konstanz (Other)
Collaborators: Université Lumière de Bujumbura (Other); The Volkswagen Foundation (Other)
Responsible Party: Principal Investigator, Anselm Crombach, Principal Investigator, University of Konstanz
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: UKULBU2014
Record Dates: First submitted 2014-09-14; First posted 2014-09-16 (Estimated); Last update posted 2017-11-29 (Actual); Status verified 2017-11

CONDITIONS: Posttraumatic Stress Disorder; Aggressive Behavior; Appetitive Aggression
Keywords: Posttraumatic Stress Disorder; Aggressive Behavior; Appetitive Aggression; Treatment; FORNET
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Aggression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- FORNET (Experimental): During FORNET, the client, with the assistance of the therapist, constructs a chronological narrative of his or her entire life with a focus on exposure to traumatic stress and committed violence. Empathic understanding, active listening, congruency and unconditional positive regard are key components of the therapist's behavior. The therapist asks in detail for the client's emotions, cognitions, physiological reactions, and sensory informations during traumatic and aggressive events to link them to an autobiographical context, namely time and place. In total the individuals receive 8 sessions of FORNET, every session lasting between 1,5 and 2 hrs depending on the needs of the participant.
  Interventions: Behavioral: FORNET
- Waiting list (No Intervention)

INTERVENTIONS:
Behavioral: FORNET
  Arms: FORNET

SUMMARY:
Soldiers deployed in peace-keeping missions as well as ex-combatants in conflict or former conflict regions were and are often exposed to multiple traumatic events and situations in which they are forced to engage in violent behavior. The treatment program Formation, Orientation and Rehabilitation by means of Narrative Exposure Therapy (FORNET) is a short-term, culturally sensitive treatment approach that aims to reduce Posttraumatic Stress Disorder (PTSD) symptoms as well as the risk to engage in uncontrolled violent behavior. Addressing trauma-related mental disorders as well as emotions related to aggression by means of FORNET is expected to facilitate reintegration in civil life and reduce uncontrolled violence.

The investigators want to provide evidence, that FORNET is an effective and efficient module to assist soldiers after deployment in Somalia and/or male and female ex-combatants who fought in the civil war in Burundi. In addition the investigators aim to explore how traumatic incidences and maltreatment during childhood may influence treatment outcomes.

ELIGIBILITY:
Inclusion Criteria:

* High degree of symptoms of posttraumatic stress disorder according to the Posttraumatic Symptom Scale,
* High degree of appetitive aggression,
* Violent behavior during the past three months

Exclusion Criteria:

* Current use of mind altering drugs,
* Psychotic symptoms

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Change in Diagnosis and load of PTSD symptoms assessed via the Posttraumatic Symptom Scale - Interview (PSS-I) | baseline, two follow-up assessments are planned within the period of 3 to 12 months post-treatment. Exact time of follow-up will be varied systematically within this period.
Change from baseline in the extend of appetitive aggression assessed via the Appetitive Aggression Scale (AAS) | baseline, two follow-up assessments are planned within the period of 3 to 12 months post-treatment. Exact time of follow-up will be varied systematically within this period.
Change in number of committed violent acts during the past three months assessed via the Domestic and Community Violence Checklist (DCVC) | baseline, two follow-up assessments are planned within the period of 3 to 12 months post-treatment. Exact time of follow-up will be varied systematically within this period.

SECONDARY OUTCOMES:
Change from baseline in load of depressive symptoms assessed via the Patient Health Questionnaire-9 (PHQ-9) | baseline, two follow-up assessments are planned within the period of 3 to 12 months post-treatment. Exact time of follow-up will be varied systematically within this period.
Change in strength of suicidal ideation measured via the Mini International Neuropsychiatric Interview (M.I.N.I.) | baseline, two follow-up assessments are planned within the period of 3 to 12 months post-treatment. Exact time of follow-up will be varied systematically within this period.
Change in physical health complains | baseline, two follow-up assessments are planned within the period of 3 to 12 months post-treatment. Exact time of follow-up will be varied systematically within this period.

CONTACTS AND LOCATIONS:
Overall Officials: Anselm Crombach, Dr., Principal Investigator — University of Konstanz
Locations (1):
- Burundian Army (FDN), Bujumbura, Burundi